CLINICAL TRIAL: NCT07260539
Title: The Effect of Education, Counseling, and Monitoring Provided to Individuals With Stoma Via a Mobile Application on Adaptation to Stoma and Quality of Lif
Brief Title: Effect of a Mobile Application on Stoma Adaptation and Quality of Life
Acronym: STOMATERAPİ-M
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ferzan Kalaycı Emek, RESEARCH ASSISTANT, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GU-HM-FKE-02; TDK-2025-10011 (Other Grant/Funding Number: Gazi University Scientific Research Projects (BAP) Coordination Unit)
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Intestinal Stoma; Ileostomy; Colostomy - Stoma
Keywords: Mobile application; ostomy; adaptation; quality of life

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two parallel groups (1:1). After baseline/pre-discharge assessment, eligible adults with a newly created intestinal stoma will be randomized using block randomization to either (A) mobile app-based education, nurse counseling, and structured monitoring plus standard care, or (B) standard care only. The trial is single-blind: participants are unaware of group assignment. Ostomy adaptation and stoma-related quality of life will be assessed at post-discharge day 15 and at months 1, 3, and 6. App usability will be assessed in Group A at month 6. All analyses will follow the intention-to-treat principle.
Who Masked: Participant
Masking Description: Participants are blinded to group allocation. The intervention is delivered by the research team, therefore care providers and investigators are not blinded. Outcomes are self-reported through digital forms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants will install the "Stomaterapi-M" mobile application on discharge day and will receive structured education (texts/videos), nurse counseling via in-app messaging and scheduled video calls, and planned monitoring for 6 months (weekly in month 1, bi-weekly in month 2, monthly in months 3-6) in addition to standard care.
  Interventions: Behavioral: Stomaterapi-M Mobile Application Support
- Standard Care (No Intervention): Participants will receive routine stomatherapy education, counseling, and follow-up provided by the clinic. Outcome assessments will be completed digitally at the same time points as the intervention group, without access to the mobile application.

INTERVENTIONS:
Behavioral: Stomaterapi-M Mobile Application Support — Participants will use the "Stomaterapi-M" mobile application for 6 months starting on discharge day. The app provides structured stoma education (texts and videos), nurse counseling via in-app messaging and scheduled video calls, and a planned monitoring module. Monitoring frequency is weekly during month 1, bi-weekly during month 2, and monthly during months 3-6, with reminder notifications before each planned entry.
  Arms: Experimental

SUMMARY:
This single-blind, parallel-group randomized controlled trial aims to evaluate the effects of a mobile app-based education, counseling, and follow-up program on stoma adaptation and quality of life in adults with a newly ostomy. The study will be conducted at the Stomatherapy Unit of Gazi University Health Research and Application Center (Ankara, Turkey). Participants meeting the inclusion criteria (n=66) will be assigned to intervention (mobile app support + standard care) and control (standard care only) groups in a 1:1 ratio via block randomization; participants will be kept unaware of their group assignment. Participants in the intervention group will download the "Stomatherapy-M" app on the day of discharge and will access structured educational content, receive nurse counseling (messaging and scheduled video calls), and share scheduled follow-up records regularly for six months. Follow-up frequency will be weekly in the first month, biweekly in the second month, and monthly in the following months. Primary outcomes; Adaptation to the stoma (Ostomy Adjustment Inventory) and stoma-related quality of life (Quality of Life Adaptation Scale) assessed at 15 days and 1, 3, and 6 months after discharge. App usability (MAUS) will be measured at 6 months only in the intervention group.

DETAILED DESCRIPTION:
This study is a single-blind, parallel-group randomized controlled trial designed to evaluate the effect of a mobile application-based education, counseling, and monitoring program on stoma adaptation and stoma-related quality of life in adults with a newly created ostomy.

The trial will be conducted at the Stomatherapy Unit of Gazi University Health Research and Application Center in Ankara, Türkiye.

Participants and sample size: Adults (≥18 years) undergoing ostomy surgery for the first time and expected to have a permanent ostomy or an ostomy lasting ≥6 months will be screened. Additional inclusion criteria include Turkish literacy, no major mental/physical/communication barriers, ownership of an iOS/Android smartphone with internet access, ability to use mobile applications, and WhatsApp use for digital form submission.

Individuals receiving concurrent stoma education/counseling from another institution or professional during follow-up will be excluded.

Based on power analysis (mixed ANOVA, Cohen f=0.40, α=0.05, power=99.7%, r=0.50), a minimum of 60 participants is required; allowing for ~10% attrition, the target enrollment is 66 participants (1:1 allocation).

Randomization and masking: Participants will be randomized 1:1 to intervention (Group A) or control (Group B) using block randomization via SealedEnvelope.com. Eleven fixed blocks of six participants will be generated, with three participants assigned to each group per block.

Randomization will be performed by an independent person not involved in data collection. The trial is single-blind: participants will not be informed of their group assignment; researchers delivering the intervention will be unblinded.

Intervention: All participants will receive the unit's standard pre-discharge stoma education and routine follow-up guidance.

In the intervention group, the "Stomaterapi-M" mobile application will be installed on discharge day with researcher guidance. For six months, participants will access structured educational materials (text and videos), nurse counseling through in-app messaging and scheduled video appointments, and a planned monitoring module for symptom/complication tracking. Monitoring frequency is weekly during month 1, bi-weekly during month 2, and monthly during months 3-6, with reminder notifications sent before each planned entry.

Participants who miss three consecutive monitoring/counseling sessions, cannot actively use the app, withdraw consent, or submit incomplete outcome forms will be removed from the study.

Control: The control group will receive standard care only, including routine stomatherapy education, counseling, and clinic follow-ups. Outcomes will be collected digitally via

Outcome measures and timeline:

Primary outcomes are (1) stoma adaptation measured with the Ostomy Adjustment Inventory (OAI), and (2) stoma-related quality of life measured with the Adaptation of Quality of Life Scale (AQLS).

These outcomes will be assessed at post-discharge day 15 and at months 1, 3, and 6.

Secondary outcome is app usability measured with the Mobile Application Usability Scale (MAUS) in the intervention group at month 6.

To minimize loss to follow-up, reminder messages/notifications will be sent to both groups at each assessment point.

Data management and analysis: Participants will be coded as A/B without linking codes to personal identifiers. Analyses will follow the intention-to-treat principle.

Group×time effects on OAI and AQLS will be analyzed using mixed two-factor repeated measures ANOVA; non-parametric equivalents will be applied if assumptions are not met. Between-group comparisons at each time point will use independent samples t-test or Mann-Whitney U test, and within-group changes will use repeated measures ANOVA or Friedman test. Significance will be set at p<0.05 (and p<0.01 where appropriate).

Ethics and funding: Ethical approval has been obtained from the Gazi University Ethics Committee (Approval No. E-77082166-302.08.01-1018511) and institutional permission from Gazi University Health Research and Application Center.

Written informed consent will be obtained from all participants. The study is funded by Gazi University Scientific Research Projects (BAP) under grant TDK-2025-10011.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years Able to read and write Turkish Undergoing ostomy surgery for the first time Permanent ostomy or expected to remain for at least 6 months No major mental, physical, or communication impairment Owns an iOS/Android smartphone with active internet access Able to use mobile applications Uses WhatsApp for digital form submission during follow-up

Exclusion Criteria:

Receiving stoma-related education or counseling from another institution or professional during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Ostomy Adjustment Inventory (OAI) Total Score | Post-discharge Day 15, Month 1, Month 3, Month 6
Adaptation of Quality of Life Scale (AQLS) Total and Subscale Scores | Post-discharge Day 15, Month 1, Month 3, and Month 6

SECONDARY OUTCOMES:
Mobile Application Usability Scale (MAUS) Score | Month 6 (intervention group only)

IPD SHARING:
Plan to Share IPD: No